CLINICAL TRIAL: NCT03153644
Title: Improving Contraceptive Care for Individuals With Chronic Conditions
Brief Title: Helping People With Health Conditions Make Birth Control Decisions
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Justine Wu, Assistant Professor, University of Michigan
Other Study IDs: HUM0012060; 1K23HD084744-01A1 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Contraception; Chronic Disease
Keywords: Qualitative Research; Medical conditions; Birth control methods; Intrauterine Devices; Physicians, Primary Care; Long-acting reversible contraceptives (LARC)
MeSH Terms: conditions — Chronic Disease | interventions — Interviews as Topic; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients: Women with chronic medical conditions
  Interventions: Behavioral: Interview
- Primary Care Providers and Medical Staff: Primary care providers can include doctors and advanced practice professionals, including midwives, nurse practitioners, and physician assistants.
  Medical staff can include social workers, nurses, medical assistants, and administrative staff
  Interventions: Behavioral: Interview
- Primary Practice: Primary care practices (family medicine, internal medicine, medicine-pediatric, or any combination of these) that at a practice-level already provide contraceptive counseling and services to reproductive-age women
  Interventions: Behavioral: Observation

INTERVENTIONS:
Behavioral: Interview — 1 hour semi-structured
  Groups: Patients; Primary Care Providers and Medical Staff
Behavioral: Observation — Field Observation
  Groups: Primary Practice

SUMMARY:
The purpose of this project is to describe how contraceptive services are currently being delivered to women with medical conditions who seek care in community-based primary care settings, such as family medicine and internal medicine clinical offices.

DETAILED DESCRIPTION:
This pilot study seeks to:

1. To understand women's beliefs, attitudes, and experiences with contraception in context of their medical conditions, drug therapy, personal preferences, and current experiences in primary care.

b. To describe provider- To describe provider- and practice-level factors that impact the delivery of contraceptive services in primary care.

To seek the perspectives of multiple stakeholders: 1) women aged 18-50 with one or more medical conditions; and 2) practice members who consist of primary care providers (PCPs) and office staff (e.g. nurses, medical assistants, and administrative staff members). The specific objective of this formative, qualitative study is to identify key patient-, provider-, and practice-level factors that are critical to the delivery of contraceptive counseling and services to women with medical conditions.

To accomplish these aims, qualitative data will be collected in clinical settings that currently provide primary care and family planning for reproductive-aged women with medical conditions. Data collected will be: 1) in-depth interviews with women with medical conditions and practice members; and 2) semi-structured observations of office activities and processes (e.g. patient check in, patient scheduling).

Using rigorous qualitative mixed methods to collect and analyze data, a deeper understanding will be gained of factors that should be considered in the design and implementation of future interventions to improve contraceptive care for women with medical conditions in primary care.

ELIGIBILITY:
Patients:

To be eligible for the study, the patient must meet all the following criteria:

* Able to speak English
* Able to give informed consent
* Have at least one significant medical condition (defined as any condition that requires medication management and/or active monitoring, like hypertension, diabetes) that would pose greater than average risk to the woman during pregnancy, including the use of medications that could be associated with potential fetal harm in the event of unplanned pregnancy (defined as medications that are Pregnancy Category C, D, or X).

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded:

* surgically or medically sterile or whose current male partner(s) are surgically or medically sterile
* females under 18 years are excluded because prior literature has shown that their healthcare and pregnancy-related experiences differ substantially enough from those of adult women.

Practice Members Inclusion Criteria:

To be eligible for the study, the practice member must meet all the following criteria:

* Age 18 or older
* Able to speak English
* Able to give informed consent
* Indirectly or directly involved with patient care

Primary Practices:

To be eligible for the study, primary care practices must meet all the following criteria:

* currently provide primary care services to reproductive-aged women aged 18-45
* currently provide prescriptions for birth control and/or provide insertion/removal of contraceptive devices (the intrauterine device or sub-dermal implant) on site OR refer patients to another site.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Identification of primary care practices (5-10) that provide primary care services and provide prescriptions for birth control and/or provide insertion/removal of contraceptive devices (the intrauterine device or sub-dermal implant) within southeast Michigan. Primary care physicians (30) and medical staff (30) within the primary care practices identified for recruitment will be approached for interviews. Approximately 30 women will be approached about participation in the study after the approval of the primary care physician. A convenience sampling approach will be used.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Factors To Guide the Design of Contraceptive Design Application | 6 months
  A semi-structured interview will be used to identify patient-, provider- and practice-level factors that are relevant to the design and implementation of a contraceptive decision aid.

CONTACTS AND LOCATIONS:
Overall Officials: Justine P WU, MD, Principal Investigator — University of Michigan
Locations (1):
- Department of Family Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Final sets of data may be shared for use via a signed Data Sharing Agreement.
  1. The organizations in the project remain the full/joint owners of such data.
  2. One of the following two conditions must be met: a. No personal health identifiers are included in the final data set; b. Appropriate patient consent and institutional review board waiver has been obtained for all identifiable data
  3. All data transferred will be in an encrypted format and stored securely.
  4. Both parties agree not to release information about specific identifiable subjects to anyone.
  5. Both parties agree to the boundary conditions of the original proposal under which data sharing was initiated.
  6. Both parties agree to support of the pertinent grant awards as part of published acknowledgments section for any document shared under this agreement.
  7. All publications arising from this shared data set must be reviewed and approved by Principle Investigator of the study.

REFERENCES:
- [Background] Chor J, Rankin K, Harwood B, Handler A. Unintended pregnancy and postpartum contraceptive use in women with and without chronic medical disease who experienced a live birth. Contraception. 2011 Jul;84(1):57-63. doi: 10.1016/j.contraception.2010.11.018. Epub 2011 Jan 20. PMID 21664511
- [Background] Naylor B. The cytologic diagnosis of cerebrospinal fluid. Acta Cytol. 1964 Mar-Apr;8(2):141-9. No abstract available. PMID 4169713
- [Background] Ornstein SM, Nietert PJ, Jenkins RG, Litvin CB. The prevalence of chronic diseases and multimorbidity in primary care practice: a PPRNet report. J Am Board Fam Med. 2013 Sep-Oct;26(5):518-24. doi: 10.3122/jabfm.2013.05.130012. PMID 24004703
- [Background] Akers AY, Gold MA, Borrero S, Santucci A, Schwarz EB. Providers' perspectives on challenges to contraceptive counseling in primary care settings. J Womens Health (Larchmt). 2010 Jun;19(6):1163-70. doi: 10.1089/jwh.2009.1735. PMID 20420508
- [Background] Dehlendorf C, Levy K, Ruskin R, Steinauer J. Health care providers' knowledge about contraceptive evidence: a barrier to quality family planning care? Contraception. 2010 Apr;81(4):292-8. doi: 10.1016/j.contraception.2009.11.006. Epub 2009 Dec 11. PMID 20227544
- [Background] Curtis KM, Tepper NK, Jamieson DJ, Marchbanks PA. Adaptation of the World Health Organization's Selected Practice Recommendations for Contraceptive Use for the United States. Contraception. 2013 May;87(5):513-6. doi: 10.1016/j.contraception.2012.08.024. Epub 2012 Oct 4. PMID 23040134
- [Background] Lee JK, Parisi SM, Akers AY, Borrero S, Schwarz EB. The impact of contraceptive counseling in primary care on contraceptive use. J Gen Intern Med. 2011 Jul;26(7):731-6. doi: 10.1007/s11606-011-1647-3. PMID 21301983
- [Background] Dicicco-Bloom B, Crabtree BF. The qualitative research interview. Med Educ. 2006 Apr;40(4):314-21. doi: 10.1111/j.1365-2929.2006.02418.x. PMID 16573666
- [Background] Crabtree BF, Miller WL. A qualitative approach to primary care research: the long interview. Fam Med. 1991 Feb;23(2):145-51. PMID 2037216
- [Derived] Wu JP, Damschroder LJ, Fetters MD, Zikmund-Fisher BJ, Crabtree BF, Hudson SV, Ruffin MT IV, Fucinari J, Kang M, Taichman LS, Creswell JW. A Web-Based Decision Tool to Improve Contraceptive Counseling for Women With Chronic Medical Conditions: Protocol For a Mixed Methods Implementation Study. JMIR Res Protoc. 2018 Apr 18;7(4):e107. doi: 10.2196/resprot.9249. PMID 29669707